CLINICAL TRIAL: NCT00153816
Title: Vitamin D/Calcium Polyp Prevention Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5R01CA098286-03 (NIH); 5R01CA098286-10 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer; Polyps; Adenomas
Keywords: Colorectal neoplasms; Adenomatous polyps
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma; Adenomatous Polyps | interventions — Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Full Factorial Placebo (Experimental): subjects in 2X2 factorial design; randomized to daily placebo
  Interventions: Drug: placebo
- Full Factorial Calcium (Experimental): subjects in 2X2 factorial design; randomized to daily 1200 mg as calcium carbonate
  Interventions: Drug: Calcium Carbonate
- Full Factorial Vitamin D (Experimental): Subjects in 2X2 factorial design; randomized to daily 1000 IU vitamin D3
  Interventions: Drug: Vitamin D3
- Full Factorial Calcium Plus Vitamin D (Experimental): Subjects in 2X2 factorial design; randomized to daily 1200 mg as calcium carbonate and 1000 IU vitamin D3
  Interventions: Drug: Calcium Carbonate; Drug: Vitamin D3
- Two Arm Placebo (Experimental): Women choosing to take daily 1200 mg as calcium carbonate randomized to daily placebo
  Interventions: Drug: Calcium Carbonate
- Two Arm Vitamin D (Experimental): Women choosing to take daily 1200 mg as calcium carbonate randomized to daily 1000 IU vitamin D3
  Interventions: Drug: Calcium Carbonate; Drug: Vitamin D3

INTERVENTIONS:
Drug: Calcium Carbonate — 3 gm/daily; 1200 mg elemental calcium/daily; two tablets per day; 600 mg elemental calcium/tablet
  Arms: Full Factorial Calcium; Full Factorial Calcium Plus Vitamin D; Two Arm Placebo; Two Arm Vitamin D
Drug: Vitamin D3 — 1000 IU/daily; two tablets per day; 500 IU per tablet
  Arms: Full Factorial Calcium Plus Vitamin D; Full Factorial Vitamin D; Two Arm Vitamin D
Drug: placebo — placebo; two tablets per day
  Arms: Full Factorial Placebo

SUMMARY:
Extensive experimental and observational data suggest that intake of calcium and of vitamin D exert protective effects on colorectal neoplasia. Building on their previous work, the investigators will investigate the chemopreventive effect of vitamin D in the large bowel, to study whether calcium with vitamin D is more effective than calcium alone, and to confirm their positive finding regarding calcium. The goal of this study is the development of chemopreventive combinations that will reduce risk of colorectal neoplasia sufficiently to permit the lengthening of surveillance intervals in most patients and to clarify important issues regarding the mechanisms of colorectal carcinogenesis and chemoprevention.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled trial of vitamin D and/or calcium supplementation for the prevention of large bowel adenomas. Subjects will be recruited from 11 Study Centers in North America. Eligible subjects will have had at least one large bowel adenoma removed in the 4 months prior to study entry and no remaining polyps in the bowel after complete colonoscopic examination. Participants will be randomized in a partial 2 x 2 factorial design to vitamin D (1000 IU/day), calcium carbonate (1200 mg elemental calcium/day), both agents, or placebo only (Full Factorial randomization). Women who decline to forego calcium supplementation will be randomized only to calcium alone or to calcium plus vitamin D (Two Arm randomization). Randomization will be stratified by gender, study center of recruitment, and anticipated follow-up interval (see below), and will be conducted separately for female subjects randomized only to vitamin D. We anticipate enrolling up to 3000 participants to reach a total of up to 2400 randomized subjects. As safety measures, blood levels of calcium, creatinine, and 25-(OH)-vitamin D will be obtained at baseline and 1 year after randomization, as well as 3 years after randomization for subjects with a 5-year surveillance cycle. Every six months after randomization subjects will complete a questionnaire regarding compliance with study agents, use of medications and vitamin/mineral supplements, illnesses, hospitalizations, and dietary intake of calcium and vitamin D. The primary endpoint of the study will be new adenomas detected on follow-up colonoscopy. These examinations are scheduled to occur either 3 years or 5 years after the qualifying examination, depending on the follow-up interval recommended by each patient's endoscopist. Some patients may, for medical reasons, have a colonoscopy at a time other than 3 or 5 years after the qualifying examination. Information from these exams will be included in analyses where appropriate. In the primary analyses, the occurrence of new adenomas in the interval between randomization and the follow-up exam will be compared between subjects randomized to vitamin D (with or without calcium) versus those randomized to no vitamin D (with or without calcium), between subjects randomized to calcium (with or without vitamin D) versus those randomized to no calcium (with or without vitamin D; excluding women electing to receive calcium who therefore cannot participate in the calcium component of the study), and between those randomized to calcium plus vitamin D versus those randomized to calcium alone. In secondary analyses, we will examine the impact of baseline vitamin D levels and vitamin D receptor (VDR) polymorphisms on the vitamin D effects. Effects on advanced adenomas will also be assessed as a secondary outcome. Participants will be invited to participate in an optional Observational Follow Up phase of the study that will begin following the end of treatment. In this phase of the study, subjects will continue to be followed on an observational basis (no study treatment) with annual questionnaires until the time of a subsequent colonoscopy that is at least three years from the follow up colonoscopy at which study treatment was ended. We will examine the occurrence of new adenomas in the interval between the colonoscopy exam at the end of study treatment and the exam at the end of observational follow up period.

ELIGIBILITY:
Inclusion Criteria:

* One or more histologically verified neoplastic polyp (adenoma) that is at least 2 mm in size removed from the large bowel with the entire large bowel examined by colonoscopy and documented to be free of further polyps or areas suspicious for neoplasia within 120 days of study entry
* Anticipated colonoscopic follow-up three years or five years after the qualifying colonoscopy
* Age between 45 and 75 years at enrollment
* (Women)Agreement to avoid pregnancy (i.e., use of standard contraception)
* Willingness to forego calcium supplementation (including multivitamins containing calcium) or, for women only, option of taking calcium supplementation of 1200 mg/daily (contained in the study pills)
* Willingness to forego vitamin D supplementation (including multivitamins containing vitamin D)
* Agreement to daily dietary intake of the equivalent of not more than 1200 mg calcium
* Agreement to daily dietary intake of the equivalent of not more than 400 IU vitamin D
* Blood calcium level within normal range
* Blood creatinine level not to exceed 20% above upper limit of normal
* Serum 25-(OH)-vitamin D within lower limit of normal to 70 ng/ml
* Ability and willingness to follow the study protocol, as indicated by provision of informed consent to participate
* Good general health, with no severely debilitating diseases or active malignancy that might compromise the patient's ability to complete the study

Exclusion Criteria:

General exclusionary criteria:

* Participation in another colorectal (bowel) study (intervention study) in the past 5 years
* Current participation in any other clinical trial (intervention study)
* Pregnancy or lactation
* A diagnosis of narcotic or alcohol dependence in the past 5 years
* A diagnosis of dementia (e.g. Alzheimer's) in the past 5 years
* A diagnosis of a significant psychiatric disability (e.g. Schizophrenia, refractory bipolar disorder, current severe depression) in the past 5 years

Exclusions due to derangement of calcium metabolism or indications /contraindications to study agents:

* Any diagnosis of kidney stones
* A diagnosis of granulomatous diseases, e.g. sarcoidosis, active chronic fungal or mycobacterial infections (tuberculosis, histoplasmosis, coccidioidomycosis, blastomycosis), berylliosis, Wegener's granulomatosis in the past 5 years
* A diagnosis of hyperparathyroidism or other serious disturbance of calcium metabolism in the past 5 years
* A diagnosis of severe kidney disease, e.g. chronic renal failure in the past 5 years
* A diagnosis of unexplained hypercalcemia in the past 5 years
* Any Diagnosis of osteoporosis with physician recommendation for treatment of low bone mass
* A diagnosis of two or more low trauma fractures in the past 5 years
* A diagnosis of a medical condition requiring treatment with vitamin D (e.g. osteomalacia) in the past 5 years

Exclusions due to intestinal or bowel problems:

* Any diagnosis of invasive carcinoma of the large bowel (even if confined to a polyp)
* Any diagnosis of familial colorectal cancer syndromes, e.g. Familial Adenomatous Polyposis (FAP) (including Gardner syndrome, Turcot's syndrome), Hereditary Nonpolyposis Colorectal Cancer (HNPCC), Hamartomatous Polyposis syndromes (including Peutz-Jeghers or Familial Juvenile Polyposis)
* Any diagnosis of inflammatory bowel disease, e.g. Crohn's Disease, Ulcerative Colitis
* A diagnosis of chronic intestinal malabsorption syndromes, e.g. celiac sprue, bacterial overgrowth, chronic pancreatitis, pancreatic insufficiency in the past 5 years
* Any large bowel resection

Exclusions due to poor health:

* A diagnosis of malignancy, other than non-melanoma skin cancer in the past 5 years
* A diagnosis of severe lung disease - class 3 or 4 (e.g. chronic obstructive pulmonary disease or emphysema requiring oxygen) in the past 5 years
* A diagnosis of severe heart disease: cardiovascular disease functional class 3 or 4 in the past 5 years
* Any diagnosis of severe liver disease, e.g. cirrhosis

Exclusions due to shipping regulations:

* Any current/past HIV positive diagnosis
* Active hepatitis B, defined as : Hep B surface antigen positive
* Active hepatitis C, defined as : measurable hepatitis C RNA

Drug exclusions:

* Use of chronic oral corticosteroid therapy in the past 5 years
* Use of lithium in the past 5 years
* Use of phenytoin's in the past 5 years
* Use of quinidine in the past 5 years
* Use of therapeutic vitamin D in the past 5 years

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2813 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Baron, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (11):
- United States (10):
  - University of Southern California, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of South Carolina, Columbia, South Carolina
  - University of Texas, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Gibbs DC, Barry EL, Fedirko V, Baron JA, Bostick RM. Impact of Common Vitamin D-Binding Protein Isoforms on Supplemental Vitamin D3 and/or Calcium Effects on Colorectal Adenoma Recurrence Risk: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2023 Apr 1;9(4):546-551. doi: 10.1001/jamaoncol.2022.6924. PMID 36701139
- [Derived] Passarelli MN, Mott LA, Barry EL, Rees JR, Baron JA. Oral Antibiotics and Risk of New Colorectal Adenomas During Surveillance Follow-up. Cancer Epidemiol Biomarkers Prev. 2021 Oct;30(10):1974-1976. doi: 10.1158/1055-9965.EPI-21-0323. Epub 2021 Jul 21. PMID 34289971
- [Derived] Passarelli MN, Karagas MR, Mott LA, Rees JR, Barry EL, Baron JA. Risk of keratinocyte carcinomas with vitamin D and calcium supplementation: a secondary analysis of a randomized clinical trial. Am J Clin Nutr. 2020 Dec 10;112(6):1532-1539. doi: 10.1093/ajcn/nqaa267. PMID 33022713
- [Derived] Crockett SD, Barry EL, Mott LA, Ahnen DJ, Robertson DJ, Anderson JC, Wallace K, Burke CA, Bresalier RS, Figueiredo JC, Snover DC, Baron JA. Calcium and vitamin D supplementation and increased risk of serrated polyps: results from a randomised clinical trial. Gut. 2019 Mar;68(3):475-486. doi: 10.1136/gutjnl-2017-315242. Epub 2018 Mar 1. PMID 29496722
- [Derived] Anderson JC, Morris CB, Robertson DJ, Barry ELR, Figueiredo JC, Cruz-Correa M, Bostick RM, Ahnen DJ, Baron JA. Can the Sum of Adenoma Diameters (Adenoma Bulk) on Index Examination Predict Risk of Metachronous Advanced Neoplasia? J Clin Gastroenterol. 2018 Aug;52(7):628-634. doi: 10.1097/MCG.0000000000000899. PMID 28767463
- [Derived] Barry EL, Peacock JL, Rees JR, Bostick RM, Robertson DJ, Bresalier RS, Baron JA. Vitamin D Receptor Genotype, Vitamin D3 Supplementation, and Risk of Colorectal Adenomas: A Randomized Clinical Trial. JAMA Oncol. 2017 May 1;3(5):628-635. doi: 10.1001/jamaoncol.2016.5917. PMID 27978548
- [Derived] Rees JR, Mott LA, Barry EL, Baron JA, Bostick RM, Figueiredo JC, Bresalier RS, Robertson DJ, Peacock JL. Lifestyle and Other Factors Explain One-Half of the Variability in the Serum 25-Hydroxyvitamin D Response to Cholecalciferol Supplementation in Healthy Adults. J Nutr. 2016 Nov;146(11):2312-2324. doi: 10.3945/jn.116.236323. Epub 2016 Sep 28. PMID 27683872
- [Derived] Rees JR, Mott LA, Barry EL, Baron JA, Figueiredo JC, Robertson DJ, Bresalier RS, Peacock JL. Randomized controlled trials: who fails run-in? Trials. 2016 Jul 29;17:374. doi: 10.1186/s13063-016-1451-9. PMID 27474021
- [Derived] Baron JA, Barry EL, Mott LA, Rees JR, Sandler RS, Snover DC, Bostick RM, Ivanova A, Cole BF, Ahnen DJ, Beck GJ, Bresalier RS, Burke CA, Church TR, Cruz-Correa M, Figueiredo JC, Goodman M, Kim AS, Robertson DJ, Rothstein R, Shaukat A, Seabrook ME, Summers RW. A Trial of Calcium and Vitamin D for the Prevention of Colorectal Adenomas. N Engl J Med. 2015 Oct 15;373(16):1519-30. doi: 10.1056/NEJMoa1500409. PMID 26465985
- [Derived] Barry EL, Mott LA, Melamed ML, Rees JR, Ivanova A, Sandler RS, Ahnen DJ, Bresalier RS, Summers RW, Bostick RM, Baron JA. Calcium supplementation increases blood creatinine concentration in a randomized controlled trial. PLoS One. 2014 Oct 15;9(10):e108094. doi: 10.1371/journal.pone.0108094. eCollection 2014. PMID 25329821
- [Derived] Barry EL, Rees JR, Peacock JL, Mott LA, Amos CI, Bostick RM, Figueiredo JC, Ahnen DJ, Bresalier RS, Burke CA, Baron JA. Genetic variants in CYP2R1, CYP24A1, and VDR modify the efficacy of vitamin D3 supplementation for increasing serum 25-hydroxyvitamin D levels in a randomized controlled trial. J Clin Endocrinol Metab. 2014 Oct;99(10):E2133-7. doi: 10.1210/jc.2014-1389. Epub 2014 Jul 29. PMID 25070320
- [Derived] Rees JR, Hendricks K, Barry EL, Peacock JL, Mott LA, Sandler RS, Bresalier RS, Goodman M, Bostick RM, Baron JA. Vitamin D3 supplementation and upper respiratory tract infections in a randomized, controlled trial. Clin Infect Dis. 2013 Nov;57(10):1384-92. doi: 10.1093/cid/cit549. Epub 2013 Sep 6. PMID 24014734
- [Derived] Bischoff-Ferrari HA, Rees JR, Grau MV, Barry E, Gui J, Baron JA. Effect of calcium supplementation on fracture risk: a double-blind randomized controlled trial. Am J Clin Nutr. 2008 Jun;87(6):1945-51. doi: 10.1093/ajcn/87.6.1945. PMID 18541589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between July 2004 and July 2008 at 11 academic medical centers and associated gastroenterology practices in the U.S.
Pre-assignment Details: 19,083 subjects were screened and 2,813 were enrolled into a run-in period of 56-84 days. 554 subjects were not randomized: 174 were ineligible due to out of range baseline lab values, 66 were ineligible for other reasons, 211 had <80% tablet adherence, and 103 refused to participate.
Period: Overall Study
Arm/Group | Full Factorial Placebo | Full Factorial Calcium | Full Factorial Vitamin D | Full Factorial Calcium Plus Vitamin D | Two Arm Placebo | Two Arm Vitamin D
Started | 415 | 419 | 420 | 421 | 295 | 289
Completed | 383 | 387 | 388 | 390 | 278 | 262
Not Completed | 32 | 32 | 32 | 31 | 17 | 27
Not completed — Death | 6 | 5 | 4 | 6 | 0 | 2
Not completed — Lost to Follow-up | 7 | 8 | 5 | 8 | 7 | 9
Not completed — Withdrawal by Subject | 9 | 9 | 9 | 4 | 1 | 5
Not completed — Follow-up exam not done | 8 | 7 | 11 | 10 | 8 | 9
Not completed — Follow-up exam done, histology missing | 2 | 3 | 3 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Factorial Placebo | Full Factorial Calcium | Full Factorial Vitamin D | Full Factorial Calcium Plus Vitamin D | Two Arm Placebo | Two Arm Vitamin D | Total
Number analyzed (Participants) | 415 | 419 | 420 | 421 | 295 | 289 | 2259
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (7.0) | 58.7 (7.0) | 58.3 (7.0) | 58.7 (6.9) | 56.7 (6.0) | 57.0 (6.6) | 58.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 63 | 62 | 67 | 295 | 289 | 836
  Male | 355 | 356 | 358 | 354 | 0 | 0 | 1423
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 24 | 26 | 28 | 26 | 146
  Not Hispanic or Latino | 395 | 395 | 396 | 394 | 267 | 263 | 2110
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 2 | 2 | 1 | 1 | 13
  Asian | 8 | 10 | 12 | 6 | 8 | 7 | 51
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 27 | 33 | 25 | 46 | 28 | 25 | 184
  White | 357 | 354 | 364 | 350 | 238 | 237 | 1900
  More than one race | 4 | 4 | 1 | 0 | 0 | 1 | 10
  Unknown or Not Reported | 13 | 15 | 16 | 17 | 20 | 18 | 99
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 7 | 7 | 7 | 7 | 5 | 4 | 37
  United States | 408 | 412 | 413 | 414 | 290 | 285 | 2222

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Adenomas
Time Frame: 1 to 10 years
Population: Subjects are included if they had a follow-up exam at least one year after randomization and had sufficient histology available to ascertain the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Factorial Placebo | Full Factorial Calcium | Full Factorial Vitamin D | Full Factorial Calcium Plus Vitamin D | Two Arm Placebo | Two Arm Vitamin D
Number analyzed (Participants) | 380 | 381 | 381 | 381 | 274 | 262
percentage of subjects | 48.2 [43.0 to 53.3] | 44.9 [39.8 to 50.0] | 47.0 [41.9 to 52.1] | 45.7 [40.6 to 50.8] | 32.1 [26.6 to 38.0] | 32.4 [26.8 to 38.5]

2. Secondary Outcome: Advanced Colorectal Lesions
Description: Includes: adenomas >=1 cm, adenomas with high grade dysplasia, adenomas with villous features, or cancer.
Time Frame: 1 to 10 years
Population: Subjects are included if they had a follow-up exam at least one year after randomization and sufficient histology available to ascertain the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Factorial Placebo | Full Factorial Calcium | Full Factorial Vitamin D | Full Factorial Calcium Plus Vitamin D | Two Arm Placebo | Two Arm Vitamin D
Number analyzed (Participants) | 380 | 386 | 384 | 387 | 276 | 261
percentage of subjects | 9.2 [6.5 to 12.6] | 11.4 [8.4 to 15.0] | 10.9 [8.0 to 14.5] | 9.6 [6.8 to 12.9] | 6.9 [4.2 to 10.5] | 7.3 [4.4 to 11.1]

ADVERSE EVENTS:
Time Frame: Events are included if they occur between randomization and 30 days after the subject exits the treatment phase of the trial, roughly 3 or 5 years after study entry, depending on when their next surveillance colonoscopy is expected.
Description: Every 6 months, subjects were asked to report all hospitalizations and contacts with medical services. All events have been confirmed via medical record review by a study physician.
Arm/Group | Full Factorial Placebo | Full Factorial Calcium | Full Factorial Vitamin D | Full Factorial Calcium Plus Vitamin D | Two Arm Placebo | Two Arm Vitamin D
Serious Adverse Events (participants affected / at risk) | 84/415 | 94/419 | 97/420 | 80/421 | 64/295 | 63/289
Other Adverse Events (participants affected / at risk) | 46/415 | 45/419 | 47/420 | 61/421 | 53/295 | 40/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Full Factorial Placebo (N=415) | Full Factorial Calcium (N=419) | Full Factorial Vitamin D (N=420) | Full Factorial Calcium Plus Vitamin D (N=421) | Two Arm Placebo (N=295) | Two Arm Vitamin D (N=289)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 1 | 0
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrhythmia (Cardiac disorders) | 4 | 3 | 4 | 3 | 1 | 3
Cardiac ischemia/myocardial infarction (Cardiac disorders) | 4 | 0 | 6 | 2 | 3 | 1
Congestive heart failure (Cardiac disorders) | 3 | 1 | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Valvular heart disease (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 0
Cochlear implant (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0
Thyroid hyperplasia (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 1 | 1
Colostomy take-down (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 0
Hiatal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ischemic colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1
Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alcohol intoxication (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Altered mental status (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Altitude sickness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 7 | 8 | 8 | 7 | 6 | 4
Deviated septum (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile Illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin hematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Multiple illnesses (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnea (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope/near syncope (General disorders) | 2 | 2 | 1 | 1 | 1 | 2
Toxic shock syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic injury (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
(General disorders) | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3 | 4 | 1 | 1 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0
Death (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Febrile Illness (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Glottitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infected prosthesis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 2 | 0 | 2
Respiratory failure (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Postoperative hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Sigmoid perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Unintentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Electrolyte disturbance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flat feet (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5 | 2 | 3 | 5
Gout/rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hernia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Joint replacement (Musculoskeletal and connective tissue disorders) | 5 | 11 | 21 | 13 | 10 | 11
Nerve entrapment (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Traumatic injury (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 1 | 0
Ventral hernia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Back pain/degenerative spinal disorders (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4 | 9 | 3 | 3
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Benign parotid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Biliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 0
Breast cancer/ductal carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/60 | 3/63 | 0/62 | 0/67 | 2 | 2 — Only women are considered at risk
Carcinoid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 1
Central nervous system cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 2
Endometrial cancer/hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/60 | 0/63 | 0/62 | 1/67 | 2 | 0 — Only women are considered at risk
Espohageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Head and neck neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0 | 0 | 1
Lymphoma/leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 1 | 0 | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0 | 0
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/60 | 0/63 | 0/62 | 0/67 | 1 | 2 — Only women are considered at risk
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Peritoneal mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Prostate and bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/355 | 1/356 | 0/358 | 0/354 | 0/0 | 0/0 — Only men are considered at risk
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12/355 | 12/356 | 13/358 | 6/354 | 0/0 | 0/0 — Only men are considered at risk
Serous ovarian tumor of low malignant potential (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/60 | 1/63 | 0/62 | 0/67 | 0 | 0 — Only women are considered at risk
Skin basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Thymoma type AB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Central nervous system cerebrovascular ischemia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cerebral spinal fluid leak (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hygroma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine syndrome (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Traumatic injury (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
(Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vertigo (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 1
Vestibular neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Bipolar affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Steroid psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cystocele/rectocele (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urolithiasis (Renal and urinary disorders) | 1 | 3 | 1 | 2 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3/355 | 5/356 | 4/358 | 1/354 | 0/0 | 0/0 — Only men are considered at risk
Breast surgery (Reproductive system and breast disorders) | 0/60 | 0/63 | 0/62 | 0/67 | 3 | 0 — Only women are considered at risk
Corpus luteum cyst (Reproductive system and breast disorders) | 0/60 | 0/63 | 0/62 | 0/67 | 1 | 0 — Only women are considered at risk
Fibroids (Reproductive system and breast disorders) | 2/60 | 0/63 | 0/62 | 0/67 | 1 | 1 — Only women are considered at risk
Pubovaginal sling (Reproductive system and breast disorders) | 0/60 | 0/63 | 0/62 | 0/67 | 1 | 0 — Only women are considered at risk
Uterine prolapse (Reproductive system and breast disorders) | 0/60 | 0/63 | 0/62 | 1/67 | 1 | 1 — Only women are considered at risk
Vaginal bleeding (Reproductive system and breast disorders) | 0/60 | 1/63 | 0/62 | 0/67 | 1 | 0 — Only women are considered at risk
Vaginal prolapse (Reproductive system and breast disorders) | 0/60 | 0/63 | 1/62 | 0/67 | 0 | 0 — Only women are considered at risk
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 3
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Traumatic injury (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cosmetic surgery (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular ischemia (Vascular disorders) | 1 | 0 | 3 | 3 | 3 | 4
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Revascularization (Vascular disorders) | 3 | 7 | 3 | 6 | 1 | 4
Subdural hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sudden death (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic injury (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Venous thromboembolism (Vascular disorders) | 1 | 2 | 6 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Full Factorial Placebo (N=415) | Full Factorial Calcium (N=419) | Full Factorial Vitamin D (N=420) | Full Factorial Calcium Plus Vitamin D (N=421) | Two Arm Placebo (N=295) | Two Arm Vitamin D (N=289)
Fracture (Musculoskeletal and connective tissue disorders) | 15 | 12 | 15 | 21 | 22 | 7
Non-melanoma skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 26 | 22 | 28 | 11 | 11
Osteopenia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 6 | 7 | 17 | 16
Hypercreatinemia (Renal and urinary disorders) | 21/407 | 29/412 | 19/415 | 29/413 | 17/294 | 9/287 — Hypercreatinemia is a value on a safety blood draw above normal for subjects whose baseline creatinine was normal. Only subjects who had at least one safety blood draw are included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No